CLINICAL TRIAL: NCT04194086
Title: Population Pharmacokinetics and Safety of Oral Posaconazole in Children With Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yang Lihua, Clinical Professor, Zhujiang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-EKZX-003
Record Dates: First submitted 2019-10-19; First posted 2019-12-11 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Leukemia, Acute
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- posaconazole as antifungal prophylaxis (Experimental)
  Interventions: Drug: posaconazole oral suspensions

INTERVENTIONS:
Drug: posaconazole oral suspensions — posaconazole oral suspensions（5mg/kg/d,tid) will be administered specially febrile neutropenia patients four times a day and blood samples will be taken any hours after the first dose at least Day 7.

SUMMARY:
This study is designed to evaluate the safety, efficacy and Population Pharmacokinetics of Oral Posaconazole in Children with leukemia.

DETAILED DESCRIPTION:
Posaconazole as a new triazole antifungal agent with broad spectrum coverage, was recommended for prophylaxis of invasive fungal disease in adults. Some studies have demonstrated the relationship between posaconazole plasma concentration and efficacy and few data have been published in children with leukemia.The purpose of this study is to describe the off-label use of posaconazole oral suspensions in children;to figure out the relationship between concentration and clinical outcomes/ adverse events;to identify factors that influence plasma concentration.

ELIGIBILITY:
Inclusion Criteria:

* 1、Patients age 2-14 years with acute leukemia (AML, ALL) undergoing chemotherapy and neutropenia expected to last at least 7 days.

  2、Karnofsky/Lansky score of 60% or greater. 3、defined as alanine transaminase (ALT) <3 x upper limit of normal (ULN),aspartate aminotransferase (AST) <3 x ULN; serum bilirubin and alkaline phosphatase <2 x ULN.

  4、No other treatment and combination of triazoles antifungals and drugs like vincristine, sirolimus, cyclosporine etc.

  5、Able to take oral medication or take medication via enteral feeding tube. 6、Ability to give informed consent. 7、No history of anaphylaxis attributed to the azole class of antifungal agents.

Exclusion Criteria:

* 1、Existing severe illness (e.g. significant cardiac, pulmonary, hepatic diseases, etc.) or major organ dysfunction.

  2、Subject is not considered eligible for this clinical research program with posaconazole.

  3、Use of medications that are known to interact with posaconazole and that may lead to life-threatening side to effects.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Number, type and grade of adverse events of posaconazole assessed by CTCAE v4.0 | 1 year
  Number, type and grade of adverse events of posaconazole oral suspensions to children with leukemia assessed by CTCAE v4.0.
Plasma posaconazole concentration monitoring and its pharmacokinetic | 1 year
  Blood samples for determination of plasma posaconazole concentration will be collected predoses (just prior to a daily dose) on days 3, 7, 14 and 21. Anther concentration (include peak concentraton) will also be collected at least 7days after the first dose.

SECONDARY OUTCOMES:
Serious Adverse events and drug-related adverse events monitoring | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No